CLINICAL TRIAL: NCT00002811
Title: A RANDOMIZED, DOUBLE BLIND, MULTI-CENTER CLINICAL STUDY TO TEST THE SAFETY AND EFFICACY OF T4N5 LIPOSOME LOTION ON PATIENTS WITH XERODERMA PIGMENTOSUM IN THE PROTECTION AGAINST ACTINIC KERATOSES
Brief Title: T4N5 Liposome Lotion Compared With Placebo Lotion for Preventing Actinic Keratoses in Patients With Xeroderma Pigmentosum
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Applied Genetics (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000064945; AGI-007; AGI-FDR000992; NCI-V96-0953
Record Dates: First submitted 1999-11-01; First posted 2004-09-02 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-05

CONDITIONS: Precancerous Condition
Keywords: actinic keratosis
MeSH Terms: conditions — Precancerous Conditions; Keratosis, Actinic | interventions — Deoxyribonuclease (Pyrimidine Dimer)

INTERVENTIONS:
Drug: liposomal T4N5 lotion

SUMMARY:
RATIONALE: Patients with xeroderma pigmentosum are more likely to develop skin lesions in sun-affected areas. These skin lesions, such as actinic keratoses, can develop into skin cancer. T4N5 liposome lotion may reduce actinic keratoses or other sun-induced skin damage in patients with xeroderma pigmentosum.

PURPOSE: Randomized double-blinded phase III trial to compare treatment using T4N5 liposome lotion with treatment using placebo in reducing actinic keratoses and other sun-induced skin damage in patients with xeroderma pigmentosum.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the safety and efficacy of T4N5 liposome lotion vs. a placebo lotion in reducing the incidence of actinic keratoses and protecting against other ultraviolet skin damage in patients with xeroderma pigmentosum.

OUTLINE: Randomized, double-blind study. Groups of 6 patients are randomly assigned in a 2:1 ratio to Arms I and II, respectively. Arm I: Chemoprevention. Lotion composed of T4 endonuclease V protein encapsulated in liposomes and suspended in phosphate-buffered saline in a hydrogel base, T4N5 Liposome Lotion, T4N5. Arm II: Control. Liposomes suspended in phosphate-buffered saline in a hydrogel base, Placebo, PLCB.

PROJECTED ACCRUAL: 6-30 patients will be entered in this multicenter study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of xeroderma pigmentosum confirmed by unscheduled DNA synthesis assay At least one histologically confirmed actinic keratosis All actinic keratoses removed prior to treatment No associated syndromes, e.g., Cockayne's syndrome or trichothiodystrophy

PATIENT CHARACTERISTICS: Age: 1.66 to 60 Other: Good general health and mental capacity No illegal drug use No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1996-07

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B. Yarosh, PhD, Study Chair — Applied Genetics
Locations (9):
- United States (7):
  - Quality Research Group, Miami Beach, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Office of Gerald Bernstein, Seattle, Washington
- Medizinische Klinik, Munich (Muenchen), Germany
- Guy's, King's and St. Thomas' Hospitals Trust, London, England, United Kingdom